CLINICAL TRIAL: NCT00066794
Title: A Phase II Study Of Induction With Daunorubicin, Cytarabine, And Cyclosporine All By Continuous IV Infusion For Previously Untreated Non-M3 Acute Myeloid Leukemia (AML) In Patients Of Age 56 Or Older
Brief Title: S0301 Cyclosporine, Daunorubicin, and Cytarabine in Treating Older Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0301; S0301 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: adult acute monocytic leukemia (M5b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); untreated adult acute myeloid leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult pure erythroid leukemia (M6b); adult erythroleukemia (M6a)
MeSH Terms: conditions — Leukemia; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities; Leukemia, Erythroblastic, Acute | interventions — Filgrastim; sargramostim; Cyclosporine; Cytarabine; Daunorubicin

INTERVENTIONS:
Biological: filgrastim — 5 mcg/kg/d IV or SC starting apx day 15
Biological: sargramostim — 250 mcg/kg/d IV or SC starting apx day 15
Drug: cyclosporine — ind: 6 mg/kg load IV over 2 hrs days 0-2 followed by 16 mg/dg/d continuous IV days 2-74 consol: 6 mg/kg load IV over 2 hrs days 0-2 followed by 16 mg/dg/d continuous IV days 2-50
Drug: cytarabine — ind: 200 mg/m2/d cont IV days 2-74
Drug: daunorubicin hydrochloride — ind: 45 mg/m2/d cont IV days 2-74

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclosporine, daunorubicin, and cytarabine, use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving cyclosporine together with daunorubicin and cytarabine works in treating older patients with untreated acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of cyclosporine, daunorubicin, and cytarabine in older patients with previously untreated acute myeloid leukemia.
* Determine the frequency and severity of toxic effects of this regimen in these patients.
* Determine, preliminarily, the frequency and prognostic significance of functional and phenotypic P-glycoprotein expression and cytogenetics in patients treated with this regimen.
* Determine, preliminarily, the pharmacokinetic characteristics of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive cyclosporine IV and daunorubicin IV continuously on days 1-3 and cytarabine IV continuously on days 1-7. Patients who achieve complete response (CR) after chemotherapy receive filgrastim (G-CSF) or sargramostim (GM-CSF) IV or subcutaneously beginning on day 15 or 20 and continuing until blood counts recover. Patients who maintain CR after 2 courses of induction therapy proceed to consolidation therapy.
* Consolidation therapy: Patients receive treatment as in induction therapy with cyclosporine and daunorubicin on days 1-2 and cytarabine on days 1-5. Patients achieving CR receive an additional course of chemotherapy beginning at least 14 days after completion of the first course of cytarabine.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 25-64 patients will be accrued for this study within 13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute myeloid leukemia (AML)

  * Differential diagnosis of AML based on FAB classification system

    * M0-M7 (No M3)
* No blastic transformation of chronic myelogenous leukemia
* Must be currently registered on protocols SWOG-9007 and SWOG-S9910

PATIENT CHARACTERISTICS:

Age

* 56 and over

Performance status

* Zubrod 0-3 (for patients 56 to 60 years of age) OR
* Zubrod 0-2 (for patients 61 to 70 years of age) OR
* Zubrod 0-1 (for patients 71 years of age and over)

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN) unless elevated unconjugated hyperbilirubinemia is secondary to Gilbert's syndrome or hemolysis and not to liver dysfunction
* AST and/or ALT no greater than 4 times ULN

Renal

* Creatinine no greater than 1.5 times ULN AND/OR
* Creatinine clearance greater than 40 mL/min

Cardiovascular

* Left ventricular function normal
* Ejection fraction at least 50% by MUGA or echocardiogram
* No unstable cardiac arrhythmias
* No unstable angina

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer that is currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent pegfilgrastim

Chemotherapy

* At least 30 days since prior low-dose cytarabine (less than 100 mg/m^2/day) for myelodysplastic syndromes and recovered
* Prior hydroxyurea to control high cell counts allowed
* No prior systemic chemotherapy for acute leukemia
* Concurrent single-dose intrathecal chemotherapy allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-07; Primary Completion 2007-02 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR) | After induction therapy is completed

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Chauncey, MD, PhD, Principal Investigator — VA Puget Sound Health Care System; Cheryl L. Willman, MD, Principal Investigator — University of New Mexico Cancer Center; Marilyn L. Slovak, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (97):
- United States (97):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Mercy Regional Cancer Center at Mercy Medical Center, Redding, California
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Tulane Cancer Center, Alexandria, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Clinic of Dr. Judy L. Schmidt, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Highland Hospital of Rochester, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming